CLINICAL TRIAL: NCT06488352
Title: Enhancing Care in Patients After Coronary Artery Bypass Graft Surgery (CABG)： OptiCABG Study
Brief Title: Enhancing Care Study in Patients After CABG
Acronym: OptiCABG
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2024-2276
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Review the data of patients who underwent coronary artery bypass grafting (CABG) at the National Center for Cardiovascular Disease, Fuwai Hospital from January 2013 to June 2023 including medical history, head CT scan, and postoperative, including 30-day mortality, arrhythmia, cerebrovascular disease and intracerebral haemorrhage, etc. Case-control and retrospective cohort studies were conducted to explore the risk factors associated with early postoperative complications, examine their relationship with postoperative management, explore independent risk factors of compound complications, and build predictive models.

ELIGIBILITY:
Inclusion Criteria:

* patients accepted CABG enrolled from January 2013 to June 2023

Exclusion Criteria:

* patients discharged within 72 hours of admission
* patients with an admission diagnosis of atrial fibrillation
* patients underwent CABG as emergency surgery
* patients underwent concurrent surgical treatments
* patients with repeat admissions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who accepted coronary artery bypass graft and met the eligibility criteria are enrolled for this study.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  The proportion of patients who die within 30 days of being admitted to the hospital.

SECONDARY OUTCOMES:
post-operative atrial fibrillation | Around the second postoperative day.
  The occurrence of atrial fibrillation after a patient has undergone surgery.
MACE | Around the second postoperative day.
  A combination of several critical cardiovascular events may vary depending on the specific context of the study or clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Structral Heart Disease Center, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No